CLINICAL TRIAL: NCT00591955
Title: Infected Elders in the Emergency Department: Outcomes and Processes of Care
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeffrey Caterino, Assistant Professor, Ohio State University
Other Study IDs: 2005H0206
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Sepsis
Keywords: geriatric; sepsis; outcome assessment(healthcare)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine factors which predict a complicated hospital course and then to develop from these findings an Emergency Department guideline to assist in knowing who is at highest risk of elderly patients with infection presenting for care.

DETAILED DESCRIPTION:
The study is looking at how closely physicians adhere to treatment guidelines in caring for elderly patients, and then to determine if there are differences in elderly patient disease symptoms that result in a failure to use guidelines. If this is known, physicians can then be aware of these differences and provide appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* blood cultures ordered in the Emergency Department
* admitted to the hospital from the Emergency Department

Exclusion Criteria:

* age less than 65
* prisoners
* Patient unable to provide consent and no legally authorized representative available
* non-English speaking
* ED visit or admission in the last 7 days for the same condition
* primary evaluation by the trauma team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 or older who present to the Emergency Department with signs that could be consistent with infection
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Complicated Clinical course | 0-30 days from ED visit
  The presense of any one of the following will constitute a complicated clinical course:
  1. mortality at 30 days
  2. requirement for ICU admission or ICU-level care withing first 48 hours
  3. positive blood cultures

SECONDARY OUTCOMES:
Inadequate process of care | entire length of Emergency Department visit and hospitalization
  failure to meet any one of the following will be considered inadequate processes of care:
  1. obtain blood cultures prior to antibiotic administration
  2. administration of antibiotics within 4 hours of presentation
  3. measure serum lactate if patient has severe sepsis in the ED
  4. Fluid resuscitation of 20-40cc/kg if mean arterial perssure is <65mmHg despite fluid resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Caterino, MD, Principal Investigator — The Ohio State University Department of Emergency Medicine
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States